CLINICAL TRIAL: NCT06645509
Title: A Phase 2, Randomised, Double-blind, Vehicle-controlled, Dose Finding, Efficacy, Tolerability and Safety Study of Victorhy in Patients With Severe Hand Hyperhidrosis
Brief Title: Severe Primary Hand Hyperhidrosis Treatment With Topical Administration of Victorhy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was early terminated due to a slower patient accrual than expected. By the expiration date of the IMP batch manufactured for the trial (30 May 2025), only 58 patients were enrolled, below the planned N of 60.
Sponsor: Dryox Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dry002-FiH; 2023-507114-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Palmar Hyperhidrosis
Keywords: Hyperhidrosis; Palmar Hyperhidrosis; Primary Palmar Hyperhidrosis; Sweat Gland Diseases; Cholinergic Antagonists
MeSH Terms: conditions — Hyperhidrosis; Sweat Gland Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding applies to Participant / Investigator & study site personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Victorhy (dose 1) (TTB gel) (Experimental): Participants will receive Victorhy (TTB, dose 1) topically to both hands, once daily for 28 days (20 participants)
  Interventions: Drug: TTB gel (dose 1)
- Victorhy (dose 2) (TTB gel) (Experimental): Participants will receive Victorhy (TTB, dose 2) topically to both hands, once daily for 28 days (20 participants)
  Interventions: Drug: TTB gel (dose 2)
- Vehicle gel (Placebo Comparator): Participants will receive a vehicle gel topically to both hands, once daily for 28 days (20 participants)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTB gel (dose 1) — A topical administration of Victorhy (TTB gel) to both hands, once daily for 28 days
  Other Names: Victorhy
  Arms: Victorhy (dose 1) (TTB gel)
Drug: TTB gel (dose 2) — A topical administration of Victorhy (TTB gel) to both hands, once daily for 28 days
  Other Names: Victorhy
  Arms: Victorhy (dose 2) (TTB gel)
Drug: Placebo — A topical administration of a vehicle (Placebo) gel to both hands, once daily for 28 days
  Arms: Vehicle gel

SUMMARY:
The objective of this study is to assess the efficacy and safety of Victorhy, a topical TTB gel in patients with severe primary hand hyperhidrosis.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, parallel group and vehicle-controlled study in which participants with severe primary hand hyperhidrosis will be randomly assigned (1:1:1) to one of the following arms:

* Victorhy dose 1
* Victorhy dose 2
* Placebo (Vehicle gel)

This study will evaluate the efficacy of Victorhy, a topical TTB gel, in patients with severe primary hand hyperhidrosis. This trial will also assess the quality of life of study participants, the rebound effect, and the pharmacokinetics of topical TTB gel. The study is intended to assess a formulation including two different doses of Victorhy (treatment groups), compared to placebo (control group) with the objective of determining the optimal therapeutic dose for use in severe hand hyperhidrosis.

Objectives:

Primary objective: To assess the efficacy of a topical TTB gel in patients with severe primary hand hyperhidrosis.

Secondary objectives:

* To assess the tolerability and safety of topical TTB gel
* To determine the optimal therapeutic dose of topical TTB gel
* To assess the quality of life of study participants
* To assess the rebound effect

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for study participation:

1. To sign an informed consent.
2. Be 18 years of age or older.
3. Be willing to comply with the study protocol.
4. Be males, or non-pregnant and non-lactating females (a negative urine pregnancy test is required for female participants of child-bearing potential).
5. Have a primary hand hyperhidrosis diagnosis for at least 6 months.
6. Have a HDSS of 3 or 4 at randomization/day 1.
7. Have a gravimetric test of at least 100 mg of sweat production at rest in each palm, and a sum of at least 250 mg in both palms, in 5 minutes (room temperature) AND/OR being on a waiting list for surgical sympathectomy.
8. Be willing to discontinue their current treatment for primary hyperhidrosis.
9. In the case of women and men of childbearing potential, for safety reasons, those who agree to follow the required contraceptive measures from the signing of the informed consent until the last study visit (day 35).

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for study participation:

1. Prior surgical procedure for hyperhidrosis.
2. Iontophoresis for the palms 4 weeks prior to randomization.
3. Treatment with botulinum toxin (e.g., Botox) for hand hyperhidrosis 6 months prior to randomization.
4. Known allergy to any of the components in the investigational product, as well as to atropine or its derivatives, e.g., ipratropium or oxitropium.
5. Subjects who are actively participating in an experimental therapy study or who received experimental therapy 30 days or 5 half-lives (whichever is longer) prior to randomization.
6. Subjects who have had a change in a regimen of psychotherapeutic medication (change in drug, dose, frequency) or who have started a psychoactive medication prior to two months of randomization.
7. Treatment with medications having systemic anticholinergic activity, centrally acting alpha-2 adrenergic agonists (e.g., clonidine, guanabenz, methyl dopa), or beta-blockers 4 weeks prior to randomization.
8. Treatment with Spiriva or similar, or any systemic treatment with an anticholinergic medication such as, but not limited to atropine belladonna, scopolamine, aclidinium, hyoscyamine, oxybutynin or glycopyrronium within 4 weeks prior to randomization.
9. Prior diagnosis of asthma or Chronic Obstructive Pulmonary Disease (COPD).
10. If female, current pregnancy or lactation.
11. Patients with skin lesions or bruisers; open wounds or inflammatory lesions on the hands or, any condition that may alter the barrier function of the skin on the hands.
12. Secondary hand hyperhidrosis or presence of a condition that may cause secondary hyperhidrosis (e.g., lymphoma, malaria, severe anxiety not controlled by medication, carcinoid syndrome, substance abuse, hyperthyroidism).
13. Known history of Sjögren's syndrome or Sicca syndrome.
14. Known history of neuromuscular disease.
15. History of glaucoma, inflammatory bowel disease, toxic megacolon, active febrile illness, paralytic ileus, unstable cardiovascular status in acute hemorrhage, severe ulcerative colitis, toxic megacolon complicating ulcerative colitis or myasthenia gravis.
16. Men with a history of urinary retention requiring catheterization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy.
17. History or presence of ventricular arrhythmias, atrial fibrillation, atrial flutter. History of other supraventricular tachycardia with a ventricular rate greater than 100 (other than sinus tachycardia).
18. Subjects who are a high medical risk because of other systemic diseases or active uncontrolled infections, or any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Mean absolute change in gravimetrically measured sweat production | From Day 1 to Day 29
Mean change in Hyperhidrosis Disease Severity Scale (HDSS) | From Day 1 to Day 29
  HDSS is a scale from grade 1 to grade 4 to measure the level of interference of sweat production with the patient's daily activities. It is the participants who give their subjective assessment, which may be:
  * Grade 1: My sweating is never noticeable and never interferes with my daily activities.
  * Grade 2: My sweating is tolerable but sometimes interferes with my daily activities.
  * Grade 3: My sweating is barely tolerable and frequently interferes with my daily activities.
  * Grade 4: My sweating is intolerable and always interferes with my daily activities.

SECONDARY OUTCOMES:
Global Impression of Change | From Day 1 to Day 29
  Overall impression of the hand sweating of the participants at day 29 compared to before treatment, ranging from 1 (much better) to 7 (much worse). It is the patients who provide their assessment of this outcome.
Proportion of participants who have an equal to or higher than 1 grade improvement in HDSS | From Day 1 to Day 29
  An improvement of 1 or more grades in the HDSS.
Proportion of participants who have an equal to or higher than 2 grade improvement in HDSS | From Day 1 to Day 29
  An improvement of 2 or more grades in the HDSS.
Proportion of participants who have at least a 50 percent reduction in gravimetrically measured sweat production | From Day 1 to Day 29
  A positive case is defined as a patient who showed a reduction of 50 percent or more in gravimetrically measured sweat production compared to day 1.
Percent change in gravimetrically-measured sweat production | From Day 1 to Day 29
  Percent change from day 1 to day 29 in the gravimetrically-measured sweat production.
Hyperhidrosis Quality of Life Index (HidroQoL) to Evaluate the Quality of Life of the Study Participants | From Day 1 to Day 29
  The HidroQoL assesses how hyperhidrosis impacts Quality of life. With 18 items on two domains, it is a comprehensive measure. The first domain with six items refers to daily life activities and the second domain with 12 items covers the psychosocial life of participants. Each item has three response options (no, not at all = 0; a little = 1; very much = 2), with a total score range from 0 to 36. The higher the score, the greater the severity. To compute scores for each dimension, items must be summed. It is the patients who provide their assessment of this outcome.
Dermatology Life Quality Index (DLQI) to Evaluate Quality of Life of Study Participants | From Day 1 to Day 29
  It consists of 10 questions referring to the past seven days. Each question of the questionnaire includes a Likert-type scale with four possible answers: "not at all", "a little", "a lot" or "very much", with scores of 0, 1, 2 and 3 respectively, with an additional option of "not relevant". The health domains included are symptoms and perceptions (questions 1, 2), daily activities (3, 4), leisure (5, 6), work/study (7), interpersonal relationships including sexuality (8, 9) and treatment (10). The sum of the scores provides a simple aggregate global value between 0 and 30, and the result can be presented as the percentage impact of the dermatologic condition on the patient's quality of life. The higher the score, the greater the impact on the patient's quality of life. It is the patients who provide their assessment of this outcome.
EQ-5D-5L Questionnaire to Evaluate the Quality of Life of the Study Participants | From Day 1 to Day 29
  It is a standardized measure of health status that provides a simple, generic measure of health. It consists of 5 items in a 5-point Likert scale and a sixth item ranged from 0 to 100. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. It is the patients who provide their assessment of this outcome.
Local skins reactions (LSRs) | From Day 1 to Day 29
  LSRs include burning/stinging, pruritus, oedema, erythema, dryness, and scaling. Each LSR will be scored as 0 (None), 1 (Mild), 2 (Moderate) or 3 (Severe). LSRs observed on a study visit day are not recorded as adverse events unless scored as 3 (Severe).
Rebound effect assessment | From Day 1 to Day 35
  To assess if on Day 35 there is an increase of 1 or more over the HDSS value obtained on Day 29 (End of Treatment Visit).

CONTACTS AND LOCATIONS:
Overall Officials: Clara Matas Nada, MD, Principal Investigator — Hospital Santa Caterina de Salt; José Gregorio Álvarez Fernández, MD, Principal Investigator — Hospital Pardo de Aravaca (Hospital Universitario Vithas Madrid Aravaca); Carmen Rodríguez Cerdeira, MD, Principal Investigator — Hospital Vithas Nosa Señora de Fátima (Hospital Vithas Vigo); Enrique Herrera Acosta, MD, Principal Investigator — Hospital Vithas Parque San Antonio (Hospital Vithas Málaga)
Locations (4):
- Spain (4):
  - Hospital Santa Caterina de Salt, Salt, Girona
  - Hospital Vithas Nosa Señora de Fátima (Hospital Vithas Vigo), Vigo, Pontevedra
  - Hospital Pardo de Aravaca (Hospital Universitario Vithas Madrid Aravaca), Madrid
  - Hospital Vithas Parque San Antonio (Hospital Vithas Málaga), Málaga